CLINICAL TRIAL: NCT04909905
Title: The Impact of Glutamine Supplementation Upon the Short-term Mortality of COVID-19 Diseased Patients Admitted in ICU: A Double Blind Randomized Clinical Trial
Brief Title: Glutamine Supplementation and Short-term Mortality in Covid-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Makram Soliman, Lecturer of anesthesia and ICU, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17300609
Record Dates: First submitted 2021-05-30; First posted 2021-06-02 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Glutamine; alanylglutamine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group EN (standard enteral nutrition) (Experimental): Patients receive standard enteral nutrition according to ICU nutrition protocol during 7days from admission
  Interventions: Dietary Supplement: Standard enteral nutrition
- Group GN (glutamine supplemented enteral nutrition) (Experimental): Patients receive intravenous glutamine supplementation to enteral nutrition in a dose of glutamine of 0.4 g/kg/day during 7 days from admission.
  Interventions: Combination Product: Glutamine

INTERVENTIONS:
Dietary Supplement: Standard enteral nutrition — Standard enteral nutrition according to ICU nutrition protocol for 7 days
  Arms: Group EN (standard enteral nutrition)
Combination Product: Glutamine — Intravenous glutamine supplementation to enteral nutrition in a dose of dose of glutamine of 0.4 g/kg/day for 7days
  Other Names: Dipeptiven
  Arms: Group GN (glutamine supplemented enteral nutrition)

SUMMARY:
The aim of this study is to investigate the effect of parenteral L-Glutamine supplementation added to enteral nutrition on short-term ICU mortality (7 days) in Covid-19 diseased patients.

DETAILED DESCRIPTION:
A written informed consent will be taken from the patients or their relatives. Patients with diagnosis of covid-19 with enteral nutrition will be enrolled. Patients will be randomly assigned to receive either standard enteral nutrition (Group EN) or intravenous glutamine supplementation to enteral nutrition (group GN) in a dose of glutamine of 0.4 g/kg/day during ICU stay.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of covid-19 diseased patients admitted to the ICU with enteral nutrition.

Exclusion Criteria:

* Renal failure (creatinine >180 mmol/l)
* Hepatic failure (bilirubin >40 mmol/l, alanine aminotransferase >100 U/l and aspartate aminotransferase >100 U/l)
* Severe neutropenia (<500 cells/mm3)
* Patients receiving cytotoxic, radiation and/or steroid therapy
* Hemodynamic instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
ICU mortality | 7 days
  Short-term ICU mortality for patients admitted in our ICU & signed for study drugs, who will expire during the study

SECONDARY OUTCOMES:
Neutrophil/lymphocyte ratio (NLR) | 7 days
  Assessing NLR at day zero & day 7 to monitor inflammatory response
D- dimer level | 7 days
  Assessing D-dimer level at day zero &day 7 to monitor coagulability status
ICU stay | 7 days
  Period of patients admission in ICU within duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Omar Soliman, MD, Principal Investigator — Omar makram
Locations (1):
- Omar Soliman, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mehta S. Nutritional status and COVID-19: an opportunity for lasting change? Clin Med (Lond). 2020 May 15;20(3):270-273. doi: 10.7861/clinmed.2020-0187. PMID 32341077